CLINICAL TRIAL: NCT05180903
Title: Clinical Performance of Polyethylene Fiber Reinforced Resin Composite Restorations (Wall Papering Technique) Versus Bulk Fill Resin Composite Restorations in Endodontically Treated Teeth: A One Year Randomized Clinical Trial
Brief Title: Clinical Performance of Polyethylene Fiber Reinforced Resin Composite Restorations (Wall Papering Technique) Versus Bulk Fill Resin Composite Restorations in Endodontically Treated Teeth Will be Evaluated Using Modified USPHS Criteria.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsattar Mohamed Metwaly, Assistant Lecturer, Conservative Department, Faculty of Dentistry., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ribbond Reinforced Composite
Record Dates: First submitted 2021-12-03; First posted 2022-01-06 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Dental Restoration Failure
Keywords: Ribbond; Reinforced Composite; polyethylene Fibers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bulk Fill resin composite restorations reinforced by ultra high molecular weight polyethylene. (Experimental): Bulk Fill resin composite restorations (X-tra base & GrandioSO, Voco, Cuxhaven, Germany) reinforced by ultra high molecular weight polyethylene. (Ribbond THM, Ribbond Inc, Seattle, WA, USA)
  Interventions: Other: X-tra base & GrandioSO reinforced by Ribbond
- Bulk Fill resin composite restorations (Active Comparator): Bulk Fill resin composite restorations (X-tra base & GrandioSO, Voco, Cuxhaven, Germany)
  Interventions: Other: X-tra base & GrandioSO reinforced by Ribbond

INTERVENTIONS:
Other: X-tra base & GrandioSO reinforced by Ribbond — The missing peripheral tooth structure will be built up via 2-mm wedge-shaped a universal hybrid resin composite, GrandioSO . Then the polyethylene fibers will be wetted with an unfilled resin first . After removing the excess resin, fibers will be covered with a very thin layer of flowable composite X-tra base . After that, fibers will be bonded immediately against the peripheral missing walls and cured for 20 seconds. Then a bulk-fill flowable resin composite lining X-tra base will be applied in approximately 4 mm thick in bulk increments as needed to fill the cavity 2 mm short of the occlusal cavosurface and each increment will be light cured for 20 s. The remaining occlusal part of the cavity will be restored with a universal hybrid resin composite, GrandioSO . The shade of the composite will be selected according to the teeth to be restored. All cavities will be restored with open-sandwich technique (Deliperi, et al. 2017).
  Other Names: Bulk Fill resin composite restorations (X-tra base & GrandioSO, Voco, Cuxhaven, Germany) reinforced by ultra high molecular weight polyethylene. (Ribbond THM, Ribbond Inc, Seattle, WA, USA)

SUMMARY:
The aim of this study will be to evaluate the clinical performance of polyethylene fiber reinforced resin composite restorations versus bulk fill resin composite restorations in endodontically treated teeth.

DETAILED DESCRIPTION:
Statement of the problem:

Restoration of non-vital teeth is always challenging for dentists. Without placing the coronal restoration, root canal treatments are not considered complete. Appropriate treatment plan selection should be based on remaining tooth structure, cavity wall thickness, tooth position in the arch, and load applied to the tooth. Previously, endodontically treated teeth (ETT) were reconstructed automatically with post, core, and full crown. But this treatment plan had many risks like root perforation, sacrificing a considerable amount of sound tooth structure, and tooth fracture.Several techniques and materials have been developed for the restoration of endodontically treated teeth including complete cast coverage, composite resins and amalgam and indirect restorations covering cusps. Resin-based materials provide rigidity and increase the fracture resistance of non-vital teeth by rein-forcing unsupported tissues. Advanced adhesive systems with improved physical properties are more aesthetic and support remaining tooth structures better than amalgam. In order to reduce polymerization shrinkage stresses, flowable resins with low elastic modulus have been suggested as a stress-absorbing layer under composite restorations. On the other hand, the use of flowable resin does not increase fracture resistance, and this layer results in contraction stresses.

Rational:

In fact, the primary aims of "biomimetic dentistry" are to be as minimally invasive as possible, and to substitute the missing hard dental tissues with restorative materials closely resembling the natural tissues regarding their mechanical features and properties.

Leno weaved Ultra-high-molecular-weight polyethylene (LWUHMWPE) fibers are plasma treated fibers. LWUHMWPE fiber reinforcement Ribbond systems (Ribbond THM, Ribbond Inc, Seattle, WA, USA) have been introduced in the attempt to increase composite resin toughness, thus increasing both durability and damage tolerance. These bondable reinforcement fibers can be closely adapted to the residual tooth structure without requiring additional preparation. The high modulus of elasticity and low flexural modulus of polyethylene fiber have a modifying effect on the interfacial stresses developed along the cavity walls.

According to a systematic review published in 2021 that was done to evaluate various in vitro studies, it was confirmed that the effect of the Ultra-high-molecular weight polyethylene fibers is increasing the fracture resistance and making more favorable fractures in endodontically treated teeth. However, there is no enough clinical data regarding this point, so this proposal is introduced.

ELIGIBILITY:
Inclusion Criteria:

Participant:

1. Patients ages 18 to 55 years.
2. Patients with endodontically treated teeth.
3. Patients with good general health.
4. Patients with good recall availability.

Teeth:

1. Successfully endotreated molar teeth.
2. Endodontically treated teeth (ETT) with at least two remaining walls.
3. ETT without apical or periapical pathosis.
4. ETT with healthy peridontium.

Exclusion Criteria:

Participant;

1. Patients who are allergic to product ingredient.
2. Patients who need indirect restorations.
3. Patients with poor oral hygiene.
4. Patients with history of bruxism and parafunctional habits.

Teeth:

1. Teeth with noncarious cervical lesions.
2. ETT with more than two remaining walls.
3. Presence of apical or periapical pathosis.
4. Teeth with advanced periodontal diseases. -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Change in the clinical performance | Change from the baseline at six months.
  Measured using modified USPHS criteria for clinical evaluation of restoration failure.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Farid Elzoghbi, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Giza, Egypt

REFERENCES:
- [Background] Abdelaziz Kandil, S. A., M. R. Farid, et al. (2021).
- [Background] Atlas A, Grandini S, Martignoni M. Evidence-based treatment planning for the restoration of endodontically treated single teeth: importance of coronal seal, post vs no post, and indirect vs direct restoration. Quintessence Int. 2019;50(10):772-781. doi: 10.3290/j.qi.a43235. PMID 31559397
- [Background] Ayna B, Celenk S, Atakul F, Uysal E. Three-year clinical evaluation of endodontically treated anterior teeth restored with a polyethylene fibre-reinforced composite. Aust Dent J. 2009 Jun;54(2):136-40. doi: 10.1111/j.1834-7819.2009.01106.x. PMID 19473155
- [Background] Durao MA, Andrade AKM, Santos MDCMDS, Montes MAJR, Monteiro GQM. Clinical Performance of Bulk-Fill Resin Composite Restorations Using the United States Public Health Service and Federation Dentaire Internationale Criteria: A 12-Month Randomized Clinical Trial. Eur J Dent. 2021 May;15(2):179-192. doi: 10.1055/s-0040-1718639. Epub 2020 Nov 26. PMID 33242913
- [Background] Deliperi S, Alleman D, Rudo D. Stress-reduced Direct Composites for the Restoration of Structurally Compromised Teeth: Fiber Design According to the "Wallpapering" Technique. Oper Dent. 2017 May/Jun;42(3):233-243. doi: 10.2341/15-289-T. PMID 28467261
- [Background] Frater M, Lassila L, Braunitzer G, Vallittu PK, Garoushi S. Fracture resistance and marginal gap formation of post-core restorations: influence of different fiber-reinforced composites. Clin Oral Investig. 2020 Jan;24(1):265-276. doi: 10.1007/s00784-019-02902-3. Epub 2019 May 16. PMID 31098711
- [Background] Garoushi S, Gargoum A, Vallittu PK, Lassila L. Short fiber-reinforced composite restorations: A review of the current literature. J Investig Clin Dent. 2018 Aug;9(3):e12330. doi: 10.1111/jicd.12330. Epub 2018 Feb 25. PMID 29479830
- [Background] Karaman E, Keskin B, Inan U. Three-year clinical evaluation of class II posterior composite restorations placed with different techniques and flowable composite linings in endodontically treated teeth. Clin Oral Investig. 2017 Mar;21(2):709-716. doi: 10.1007/s00784-016-1940-y. Epub 2016 Aug 19. PMID 27538739
- [Background] Kashi, A. M. A., S. Ghanbaran, et al. (2020).
- [Background] Lempel E, Lovasz BV, Bihari E, Krajczar K, Jeges S, Toth A, Szalma J. Long-term clinical evaluation of direct resin composite restorations in vital vs. endodontically treated posterior teeth - Retrospective study up to 13 years. Dent Mater. 2019 Sep;35(9):1308-1318. doi: 10.1016/j.dental.2019.06.002. Epub 2019 Jul 2. PMID 31278018
- [Background] Ozsevik AS, Yildirim C, Aydin U, Culha E, Surmelioglu D. Effect of fibre-reinforced composite on the fracture resistance of endodontically treated teeth. Aust Endod J. 2016 Aug;42(2):82-7. doi: 10.1111/aej.12136. Epub 2015 Nov 27. PMID 26611674
- [Background] Shah EH, Shetty P, Aggarwal S, Sawant S, Shinde R, Bhol R. Effect of fibre-reinforced composite as a post-obturation restorative material on fracture resistance of endodontically treated teeth: A systematic review. Saudi Dent J. 2021 Nov;33(7):363-369. doi: 10.1016/j.sdentj.2021.07.006. Epub 2021 Jul 14. PMID 34803275
- [Background] Valizadeh S, Ranjbar Omrani L, Deliperi S, Sadeghi Mahounak F. Restoration of a Nonvital Tooth with Fiber Reinforce Composite (Wallpapering Technique). Case Rep Dent. 2020 Jun 5;2020:9619787. doi: 10.1155/2020/9619787. eCollection 2020. PMID 32566326
- [Background] Wang X, Shu X, Zhang Y, Yang B, Jian Y, Zhao K. Evaluation of fiber posts vs metal posts for restoring severely damaged endodontically treated teeth: a systematic review and meta-analysis. Quintessence Int. 2019;50(1):8-20. doi: 10.3290/j.qi.a41499. PMID 30600326
- [Derived] Metwaly AA, Elzoghby AF, Abd ElAziz RH. Clinical performance of polyethylenefiber reinforced resin composite restorations in endodontically treated teeth: (a randomized controlled clinical trial). BMC Oral Health. 2024 Oct 24;24(1):1285. doi: 10.1186/s12903-024-05009-8. PMID 39448991